CLINICAL TRIAL: NCT01662050
Title: Phase II Study of Age-Adjusted R-BAC (Rituximab, Bendamustine, Cytarabine) as Induction Therapy in Older Patients With Mantle Cell Lymphoma (MCL)
Brief Title: Phase II Study of Age-Adjusted Rituximab, Bendamustine, Cytarabine as Induction Therapy in Older Patients With MCL
Acronym: FIL-RBAC500
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL-RBAC500
Record Dates: First submitted 2012-06-26; First posted 2012-08-10 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: MCL; Mantle Cell Lymphoma; Older
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Bendamustine Hydrochloride; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One arm for all patients. (Experimental): Rituximab, Bendamustine, Cytarabine
  Interventions: Drug: Rituximab, Bendamustine, Cytarabine.

INTERVENTIONS:
Drug: Rituximab, Bendamustine, Cytarabine. — 6 cycles of 28 days with Rituximab, Bendamustine and Cytarabine (R-BAC). Rituximab 375mg/mq; Bendamustine 70mg/mq; Cytarabine 500mg/mq.

SUMMARY:
A phase 2 study of standard R-BAC (rituximab 375 mg/m2, bendamustine 70 mg/m2, ara-c 800 mg/m2) has been recently ultimated at the Vicenza Hematology Department involving several regional centers on both untreated and previously treated patients with Mantle Cell Lymphoma (MCL). An interim analysis conducted on 30 patients showed that rituximab + bendamustine + ara-c combination had very good clinical activity, but a quite relevant hematological toxicity, especially in previously treated and older patients (Visco C, ICML 2011 Lugano Conference, Poster 236).

Objectives:

The primary objective is to determine the activity (complete remission rate according to Cheson 2007 criteria) and safety of age-adjusted Rituximab-Bendamustine-Cytarabine (RBAC500) regimen at the end of treatment in older untreated patients with MCL.

The secondary objectives are to determine:

* The rate of molecular response (characterized by labs of the FIL)
* The progression-free survival (PFS)
* The overall survival (OS)
* The duration of responses (DOR)
* The rate of patients that complete the expected treatment schedule (6 courses)
* The rate of patients that are subject to dose reductions or delays

DETAILED DESCRIPTION:
Study End points Primary efficacy end point of the study is the proportion of CR defined according to Cheson criteria (2007) at the end of treatment (6 or 4 cycles). Primary safety end point is the occurrence of any of the stop treatment criteria or of any episode of relevant toxicity, as above defined.

Secondary end points are MRD defined response, OS, PFS and DOR (Cheson 2007). Molecular response is the proportion of patients with molecular rearrangements at baseline that become negative during treatment, measured by qualitative and quantitative PCR.

OS is measured from enrollment until death from any cause. PFS is measured from the time of enrollment until disease progression, relapse or death from any cause. DOR is measured from the first assessment that documents response (CR or PR) to the date of disease relapse or progression. Minimum follow up required for all patients will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with MCL aged > 65 years if they are FIT according to the geriatric CGA assessment.
* age 60-65 years not eligible to high-dose chemotherapy plus transplantation, FIT or UNFIT according to the geriatric CGA assessment.
* ECOG performance status ≤ 2.
* Positivity for cyclin D1 and SOX11 [the latter being mandatory in cases lacking cyclin D1- or t(11;14)-negative], CD20 and CD5.
* Adequate renal function (Creatinine clearance > 40 mL/min), with preserved diuresis.
* Adequate liver function: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN) value, total bilirubin < 2 mg/dL, unless directly attributable to the patient's tumor.
* Hepatitis B core antibody (HBcAb) positive/HBsAg negative/HBV-DNA negative patients may be enrolled if correct antiviral prophylaxis is administered at least 2 weeks before initiating protocol treatment.
* Written informed consent.

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive.
* Previous treatment for lymphoma
* Medical conditions or organ injuries that could interfere with administration of therapy.
* Active bacterial, viral, or fungal infection requiring systemic therapy.
* Seizure disorders requiring anticonvulsant therapy.
* Severe chronic obstructive pulmonary disease with hypoxemia.
* History of severe cardiac disease: New York Heart Association (NYHA) functional class III-IV, myocardial infarction within 6 months, ventricular tachyarrhythmias, dilatative cardiomyopathy, or unstable angina.
* Uncontrolled diabetes mellitus.
* Active secondary malignancy.
* Known hypersensitivity or anaphylactic reactions to murine antibodies and proteins, to Bendamustine or mannitol.
* Major surgery within 4 weeks of study Day 1.
* HBsAg+
* HCVAb+ patients with active viral replication (HCV-RNA+ with AST > 2 x normal limit)
* Any co-existing medical or psychological condition that would preclude participation in the study or compromise the patient's ability to give informed consent, or that may affect the interpretation of the results, or render the patient at high risk from treatment complications.
* CNS involvement (a diagnostic lumbar puncture will be performed in patients with the blastoid variant of MCL)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-03-20 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
complete remission rate at the end of treatment | 6 months
  The primary objective is to determine the activity [complete remission rate (CR) according to Cheson 2007 criteria]
Toxicity will be represented by the occurrence of any of the stop treatment criteria or of any episode of relevant toxicity | 6 months
  Relevant toxicity:
  Grade 4 cytopenia lasting for more than 6 days or Grade 3-4 non-hematologic toxicity or Febrile neutropenia lasting for more than 3 consecutive days.
  Stop treatment criteria:
  1. Occurrence of relevant toxicity for two subsequent or consecutive cycles.
  2. Grade 3-4 hematological or non-hematological toxicity on day +28 of a cycle not resolving within two weeks.
  3. Grade 3-4 hematological or non-hematological toxicity on day +28 of a cycle after 25% dose reduction.
  4. Patient refusal to procede with further cycles due to perceived excessive toxicity.
  5. Any unpredictable drug related event that suggests against study continuation

SECONDARY OUTCOMES:
the rate of molecular response | 6 months
  the rate of molecular response (characterized by labs of the FIL)
the progression-free survival (PFS) | 30 months
  the progression-free survival (PFS)is defined as the time from enrollment to complete remission with disappearance of all evidence of disease, disease progression or relapse or death from any cause.
the overall survival (OS) | 30 months
  the overall survival (OS) is defined as the time from enrollment to death from any cause
the duration of responses (DOR) | 30 months
  the duration of responses (DOR)
the rate of completion of treatment | 6 months
  the rate of patients that complete the expected treatment schedule (6 courses)
the rate of dose reductions or delays | 6 months
  the rate of patients that are subject to dose reductions or delays

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Visco, MD, Principal Investigator — Ospedale ULSS 6 di Vicenza - Ematologia
Locations (56):
- Italy (56):
  - A.O. Policlinico Consorziale, Bari, BA
  - IRCCS Ospedale Oncologico, Bari, BA
  - A.O. Spedali Civili, Brescia, BS
  - U.O.C. Ematologia Ospedale "San Nicola Pellegrino" ASL BAT, Trani, BT
  - Ospedale Businco, Cagliari, CA
  - AO Valduce, Como, CO
  - U.O.C. Garibaldi Nesima, Catania, CT
  - AOU Careggi, Florence, FI
  - A.O.U. San Martino, Genova, GE
  - PO Vito Fazzi, Lecce, LE
  - Ospedale Cardinale G. Panico, Tricase, LE
  - Asur - Zona Territoriale 8, Civitanova Marche, MC
  - U.O.C. Ematologia - Policlinico Universitario, Messina, ME
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - A.O. S. Carlo Borromeo di Milano Unità Semplice di Trapianto Midollo - A.O.S.Carlo Borromeo, Milan, MI
  - A.O. Niguarda, Milan, MI
  - Osp. San Gerardo, Monza, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Centro Oncologico Modenese (COM), Modena, MO
  - "La Maddalena", Palermo, PA
  - Ospedali Riuniti Villa Sofia - Cervello, Palermo, PA
  - Ospedale Civile Guglielmo da Saliceto, Piacenza, PC
  - Università di Padova, Padua, PD
  - Presidio ospedaliero di Pescara, Pescara, PE
  - CRO Aviano, Aviano, PN
  - Fondazione IRCCS Policlinico San Matteo,, Pavia, PV
  - Osp. S. Maria delle Croci, Ravenna, RA
  - Azienda Ospedaliera "Bianchi Melacrino Morelli", Reggio Calabria, RC
  - Azienda Ospedaliera Arcispedale "S.Maria Nuova", Reggio Emilia, RE
  - A.O. San Camillo Forlanini, Roma, RM
  - Nuovo Regina Margherita, Roma, RM
  - Università "La Sapienza", Roma, RM
  - A.O. S. Giovanni Addolorata, Roma, RM
  - Ospedale degli Infermi di Rimini, Rimini, RN
  - Azienda ULSS 18, Rovigo, RO
  - Osp. Umberto I, Nocera Inferiore, SA
  - A.O.U. San Giovanni di Dio e Ruggi d'Aragona, Salerno, SA
  - Az. Ospedaliera Univ. Senese, Siena, SI
  - ASL TO4, Ciriè-Ivrea-Chivasso, TO
  - Ospedale S. Luigi Gonzaga,, Orbassano, TO
  - A.O.U. S. Giovanni Battista -Ematologia 2, Torino, TO
  - AOU San Giovanni Battista-Ematologia 1, Torino, TO
  - A.O. S. Maria di Terni, Terni, TR
  - Azienda Ospedaliero - Universitaria di Udine, Udine, UD
  - Ospedale di Circolo e Fondazione Macchi - Ematologia, Varese, VA
  - Ospedale di Circolo e Fondazione Macchi - Oncologia, Varese, VA
  - Osp. S. Andrea Vercelli, Vercelli, VC
  - Ospedale Civile di Mirano, Mirano, VE
  - Ospedale San Bortolo, Vicenza, VI
  - Ospedale Policlinico G.B. Rossi (Borgo Roma) Di Verona, Verona, VR
  - A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Comprensorio sanitario di Bolzano, Bolzano
  - Ospedale Cardarelli, Campobasso
  - A.O. Pugliese-Ciacci, Catanzaro
  - IRST, Meldola
  - Università del Piemonte Orientale - Novara, Novara

REFERENCES:
- [Derived] Tisi MC, Moia R, Patti C, Evangelista A, Ferrero S, Spina M, Tani M, Botto B, Celli M, Puccini B, Cencini E, Di Rocco A, Chini C, Ghiggi C, Zambello R, Zanni M, Sciarra R, Bruna R, Ferrante M, Pileri SA, Quaglia FM, Stelitano C, Re A, Volpetti S, Zilioli VR, Arcari A, Merli F, Visco C. Long-term follow-up of rituximab plus bendamustine and cytarabine in older patients with newly diagnosed MCL. Blood Adv. 2023 Aug 8;7(15):3916-3924. doi: 10.1182/bloodadvances.2023009744. PMID 37171620
- [Derived] Visco C, Chiappella A, Nassi L, Patti C, Ferrero S, Barbero D, Evangelista A, Spina M, Molinari A, Rigacci L, Tani M, Rocco AD, Pinotti G, Fabbri A, Zambello R, Finotto S, Gotti M, Carella AM, Salvi F, Pileri SA, Ladetto M, Ciccone G, Gaidano G, Ruggeri M, Martelli M, Vitolo U. Rituximab, bendamustine, and low-dose cytarabine as induction therapy in elderly patients with mantle cell lymphoma: a multicentre, phase 2 trial from Fondazione Italiana Linfomi. Lancet Haematol. 2017 Jan;4(1):e15-e23. doi: 10.1016/S2352-3026(16)30185-5. Epub 2016 Dec 5. PMID 27927586